CLINICAL TRIAL: NCT03086421
Title: Social Emotional Development in Young Children With Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: SEDYC; NCI-2021-05585 (Registry Identifier: NCI)
Record Dates: First submitted 2017-03-10; First posted 2017-03-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor, Childhood; Brain Tumor, Pediatric
Keywords: Childhood cancer; Social functioning; Social development
MeSH Terms: conditions — Brain Neoplasms; Neoplasms; Social Adjustment | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Brain Tumor Participants: Participants with a diagnosis of brain tumor who are between the ages of 4 and 6 years old and are 6 to 12 months post-completion of treatment. They will complete several standard questionnaires.
  Interventions: Behavioral: Questionnaires
- Solid Tumor Participants: Participants with a diagnosis of non-Central Nervous System (non-CNS) solid tumor who are between the ages of 4 and 6 years old and are 6 to 12 months post-completion of treatment. They will complete several standard questionnaires.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Participants, their parent/legal guardian, and if consented to another adult caregiver will be asked to complete several questionnaires evaluating the participant's social cognitive skills, social experience, neurocognitive functioning, and neurocognitive skills.
  Other Names: Psychological Evaluation; Standardized Testing

SUMMARY:
Many children with cancer are diagnosed in early childhood, and as such, will likely miss key social experiences such as participation in preschool or kindergarten, playing on playgrounds, and other normative experiences. In typically-developing children, it is known that these experiences - and the skills that are learned during them - are critical to later well-being. Very little is known about the psychological functioning of young children with cancer, as studies have predominantly focused on those who are older (at least 8 years of age). This study will explicitly assess social functioning in preschool-aged children with cancer and follow the development of their social functioning from the end of treatment into survivorship.

The goals of this pilot study are to begin to assess the impact of missed early childhood social experiences, as well as the interaction with developing neurocognitive problems.

PRIMARY OBJECTIVE: Explore the impact of cancer in the central nervous system on social functioning of young children (ages 4-6) after completion of therapy.

DETAILED DESCRIPTION:
Participants will be evaluated using the same or similar questionnaires at two time points. The first assessment will take place when they are 6-12 months post the end of treatment. Participants and their parents/legal guardian will complete an assessment of social and cognitive functioning by completing questionnaires about social, emotional, behavioral, and executive functioning. If the study participant agrees, they will identify another adult (that is, teacher or daycare employee) who may be contacted to complete questionnaires about the participant's social and behavioral functioning. A follow-up study visit will occur about two years later.

ELIGIBILITY:
Inclusion Criteria:

* Primary Diagnosis of a brain or non-CNS solid tumor
* Between 4 and 6 years of age at enrollment
* Between 6 and 12 months post-therapy at the time of enrollment
* Treatment plan included chemotherapy
* English speaking
* Cognitive and language capacity to complete measures

Exclusion Criteria:

* Diagnosis of a genetic disorder/pre-existing neurodevelopmental condition associated with neurocognitive or social impairment (e.g., autism, Neurofibromatosis Type 1 (NF1), Down syndrome)
* Solid tumor patients who required CNS-directed therapy (e.g., radiation, intrathecal chemotherapy)
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be patients at St. Jude Children's Research Hospital who meet the eligibility criteria, along with their parent/legal guardian, and another adult caregiver.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Social functioning as assessed by parent-completed measures and child-completed measures | All measures will be completed at both the study enrollment and 24±3 months later
  Descriptive statistics will be provided. Parents will complete the Social Competence Inventory, Quality of Play Questionnaire, and the NIH Toolbox. Patients completed measures include the subtests from the NIH Toolbox, Challenging Situations Task, and Developmental Neuropsychological Assessment (2nd edition). Analyses will be completed to assess performance on these measures at each time point and to assess change over time. Analyses will be completed by diagnostic group (brain tumor versus solid tumor).

CONTACTS AND LOCATIONS:
Overall Officials: Heather Conklin, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

DOCUMENTS (1):
  • Informed Consent Form (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT03086421/ICF_000.pdf